CLINICAL TRIAL: NCT00175045
Title: A Phase 2, Open-Label Multicenter Study to Evaluate the Pharmacodynamics of Intravenous Lansoprazole to That of Oral Lansoprazole in Subjects With Erosive Esophagitis
Brief Title: Intravenous vs Oral Lansoprazole on Gastric Acid Secretion in Subjects With Erosive Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP Clinical Sciences, Takeda Global Research & Development Center, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C02-039; U1111-1114-2148 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Esophagitis; Reflux
Keywords: Intravenous; gastric acid secretion; Lansoprazole; Esophagitis; reflux
MeSH Terms: conditions — Esophagitis; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole IV 30 mg QD (Experimental)
  Interventions: Drug: Lansoprazole
- Lansoprazole Capsule 30 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 30 mg, intravenous injection, once daily for up to 7 days.
  Arms: Lansoprazole IV 30 mg QD
Drug: Lansoprazole — Lansoprazole 30 mg, capsules, orally, once daily for up to 7 days.
  Other Names: AG-1749
  Arms: Lansoprazole Capsule 30 mg QD

SUMMARY:
The purpose of this study was to compare the pharmacodynamics of intravenous (IV) lansoprazole to oral lansoprazole capsules, once daily (QD), in participants with erosive esophagitis.

DETAILED DESCRIPTION:
Phase 2, open label, multi-center, 2-period study to compare the pharmacodynamics of IV lansoprazole 30 mg to oral lansoprazole 30 mg in subjects with erosive esophagitis (grade >or= 2)diagnosed by endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were required to have Grade 2, 3 or 4 esophageal findings according to the TAP Grading Scale during the pretreatment endoscopy.
* Subjects must discontinue histamine H2-receptor antagonists, proton pump ® inhibitors, prokinetic agents, antacids and Carafate before the first dose of drug and during the study.

Exclusion Criteria:

* Gastric or duodenal ulcer (a lesion with appreciable depth ≥3 mm) or a hiatal hernia >5 cm.
* Subjects could not have a diagnosis of Barrett's esophagus (with or without dysplastic changes).
* Co-existing systemic disease affecting the esophagus, (ie, scleroderma, viral or fungal infection), radiation therapy to the region of the esophagus, or caustic or physiochemical trauma to the esophagus.
* Current esophageal stricture requiring dilatation. The endoscope had to pass freely into the stomach during endoscopy. Any strictures could not have been dilated within 12 weeks before beginning the Pretreatment Period.
* Positive H pylori by rapid urease test (CLO® test Kimberly-Clark Corporation).
* Uncontrolled, clinically significant cardiovascular, pulmonary, renal, hepatic, metabolic, gastrointestinal, neurological or endocrine disease or other abnormality (other than the erosive esophagitis disease being studied).
* Diagnosis of Zollinger-Ellison syndrome, esophageal varices, symptomatic pancreaticobiliary tract disease, cholecystitis, rheumatoid arthritis, lupus, or malignancy (except basal cell carcinoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-06; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Maximal Acid Output obtained 22 hours after the last dose of IV lansoprazole compared to the Maximal Acid Output obtained 22 hours after the last dose of oral lansoprazole following pentagastrin stimulation in both instances. | Day 7 vs Day 15

SECONDARY OUTCOMES:
Basal Acid Output obtained 21 hours after the last dose of IV lansoprazole compared with that obtained 21 hours after the last dose of oral lansoprazole. | Day 7 vs Day 15
Maximum Acid Output and Basal Acid Output measurements obtained 21 hours and 22 hours, respectively, after the first dose of IV lansoprazole versus those obtained after the last dose of oral lansoprazole. | Day 7 vs Day 8
Maximum Acid Output and Basal Acid Output results obtained after the first versus last dose of IV lansoprazole. | Day 8 vs Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda